CLINICAL TRIAL: NCT04379908
Title: Healthy Lifestyles and Quality of Life in Women With Breast Cancer (Health-EpiGEICAM)
Brief Title: Healthy Lifestyles and Quality of Life in Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Asociación Española contra el Cáncer (Other)
Responsible Party: Sponsor
Other Study IDs: Health-EpiGEICAM
Record Dates: First submitted 2020-04-29; First posted 2020-05-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Lifestyle; Quality of life; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Samples of stored primary tumor tissue will be collected (if available) in order to obtain high-quality molecular data to gain a better understanding of breast cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional, multicenter, and observational study designed to update clinical, pathological, and lifestyle information for a cohort of approximately 1245 breast cancer patients included in the epiGEICAM-01 study.

DETAILED DESCRIPTION:
In 2007, GEICAM started the EpiGEICAM case-control study, to investigate the association of diet and other lifestyle factors with breast cancer risk. In this study, we were able to identify two dietary patterns related with breast cancer in an opposite way. Thus, while women with high adherence to the so-called "Western" diet had an excess risk of breast cancer, high adherence to the "Mediterranean" pattern reduced the risk of breast cancer, being this effect particularly marked for triple negative tumors. Regarding physical activity, our preliminary results show a positive association between sedentarism and breast cancer risk. This project will focus on breast cancer patients included in that study in order to explore their degree of adherence to lifestyle behaviour recommendations and their association with the quality of life of these women.

Survivors will be re-surveyed to assess tobacco, alcohol, diet, obesity and health-related quality of life, using a specific questionnaire witch contains the following information:

* Sociodemographic information.
* Anthropometric data (weight, height).
* Clinical and gynecological data.
* Assessment of lifestyle habits: including tobacco consumption and diet.
* Physical activity questionnaire, with the International Physical Activity Questionnaire (IPAQ).
* Questionnaire to know the preference of patients on receiving information about their treatment in physical exercise.
* General Short Form-36 (SF36) quality of life questionnaire already used at the time of diagnosis.
* Specific Fatigue and Quality of Life Questionnaires: Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) and Functional Assessment of Cancer Therapy - Fatigue (FACT-F).
* Coping questionnaires: COPE-28 and Brief Resilience Scale (BRS).

ELIGIBILITY:
Inclusion Criteria:

* Women who participated in the case cohort in the epiGEICAM-01 clinical epidemiological study
* Capable and willing women to provide their written informed consent. If the patient has died, the biological sample and clinical data may be analyzed in those cases in which there is no express opposition from the patient or her relatives for participation in this type of study. The document of previous instructions will be consulted and, failing that, the criteria of the closest relative of the deceased will be recorded.
* Capable and willing women to complete the questionnaires provided in the study (except deceased).

Exclusion Criteria: None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer who have previously participated in the epiGEICAM-01 study.
Sampling Method: Non-Probability Sample
Enrollment: 801 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Degree of adherence of breast cancer survivors to international guidelines regarding modifiable lifestyles by questionnaires | After completing the survey, an average of 1 week
  The scores that measure the degree of compliance with the World Cancer Research Fund (WCRF) / American Institute for Cancer Research (AICR) recommendations and those included in the European Code Against Cancer 4th edition (CECC4) at the time of diagnosis (time 1) and those obtained in the second interview (time 2) will be calculated and described. Differences will be described using basic descriptive statistics and the statistical significance of the differences found using the paired samples hypothesis contrast test (repeated measurements on the same woman). To assess which factors are associated with changes in the degree of compliance, repeated measures mixed models will be used, considering each woman as a term with random effects.
  The specific questionnaires that will be used are Anthropometric data, Assessment of lifestyle habits, International Physical Activity Questionnaire (IPAQ).
Quantify changes in modifiable lifestyles by questionnaires | After completing the survey, an average of 1 week
  The scores that measure the degree of compliance with the World Cancer Research Fund (WCRF) / American Institute for Cancer Research (AICR) recommendations and those included in the European Code Against Cancer 4th edition (CECC4) at the time of diagnosis (time 1) and those obtained in the second interview (time 2) will be calculated and described. Differences will be described using basic descriptive statistics and the statistical significance of the differences found using the paired samples hypothesis contrast test (repeated measurements on the same woman). To assess which factors are associated with changes in the degree of compliance, repeated measures mixed models will be used, considering each woman as a term with random effects.
  The specific questionnaire that will be used is Assessment of lifestyle habits
Differences in adherence to recommendations of survivors of breast cancer | After completing the survey, an average of 1 week
  The scores that measure the degree of compliance with the World Cancer Research Fund (WCRF) / American Institute for Cancer Research (AICR) recommendations and those included in the European Code Against Cancer 4th edition (CECC4) at the time of diagnosis (time 1) and those obtained in the second interview (time 2) will be calculated and described. Differences will be described using basic descriptive statistics and the statistical significance of the differences found using the paired samples hypothesis contrast test (repeated measurements on the same woman). To assess which factors are associated with changes in the degree of compliance, repeated measures mixed models will be used, considering each woman as a term with random effects.
  The specific questionnaires that will be used are Sociodemographic information, Clinical and gynecological data and Coping questionnaires: COPE-28 and Brief Resilience Scale (BRS).
Estimate the health-related quality of life (HRQL) of these patients in all its dimensions and compare it with that observed in the general population and with the self-reported by these women at the time of diagnosis | After completing the survey, an average of 1 week
  The HRQL will be estimated at the present time and at diagnosis, computing the Short Form-36 Health Survey scores in the 8 dimensions included in the questionnaire and the two summarizing components. To compare the HRQL observed in these women with those of the Spanish population, standardized values of these dimensions will be used, considering the mean and standard deviation observed in the general population. The Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) and the Functional Assessment of Cancer Therapy - Fatigue (FACT-F) questionnaire will be assessed according to the FACT scoring standards.
  The higher the number of points, the better the quality of life. To obtain the score, the negative questions are reverted; then the answers of the domains are added up, and a proportional average is carried out in case of non answered items.
Adherence effect to the WCRF, AICR and CECC4 recommendations on the HRQL | After completing the survey, an average of 1 week
  Adherence effect to recommendations (measuring each of them separately and global adherence) has a positive impact on the HRQL of these women.
  Global adherence score to the WCRF / AICR recommendations and to those included in the CECC4 on each of the HRQL dimensions will be quantified, using multiple regression models including age adjustment variables, the time from diagnosis, stage, situation with respect to the tumor (without disease or with disease) and socioeconomic status, as well as all those that act as confounding factors (those that are associated with HRQL and the degree of adherence to the recommendations ). Outcome variable: HRQL dimensions; Main exposure variable: Index of compliance with the recommendations.
  The specific questionnaires that will be used are General Short Form-36 quality of life questionnaire, Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) and Functional Assessment of Cancer Therapy - Fatigue (FACT-F).
Compliance effect to the WCRF, AICR and CECC4 recommendations on survival of these women. | After completing the survey, an average of 1 week
  Cox regression models will be used to explore the influence that initial adherence to these recommendations has had on disease-free survival and overall survival for these women. Result variable: Time until the occurrence of the event / censorship; Main exposure variable: Degree of initial compliance with the recommendations.
  Disease-free survival is defined as the time from initially diagnosis to the first documented progression disease, or death from any cause, whichever occurs first.
  Overall survival is defined as the time from the date of initially diagnosis to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Instituto de Salud Carlos III; Study Director, Study Director — Hospital General Universitario Gregorio Marañón
Locations (18):
- Spain (18):
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, Galicia
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Centro Oncológico de Galicia, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Virgen de los Lirios, Alicante
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Puerta del Mar, Cadiz
  - ICO de Girona, Hospital Dr. Josep Trueta, Girona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Lope V, Guerrero-Zotano A, Ruiz-Moreno E, Bermejo B, Antolin S, Montano A, Baena-Canada JM, Ramos Vazquez M, Fernandez de Larrea-Baz N, Chacon JI, Garcia-Saenz JA, Olier C, Munoz M, Anton A, Sanchez Rovira P, Arcusa Lanza A, Gonzalez S, Oltra A, Brunet J, Gavila Gregori J, Martinez MT, Calvo L, Rosell L, Bezares S, Pastor-Barriuso R, Perez-Gomez B, Martin M, Pollan M. Clinical and Sociodemographic Determinants of Adherence to World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) Recommendations in Breast Cancer Survivors-Health-EpiGEICAM Study. Cancers (Basel). 2022 Sep 27;14(19):4705. doi: 10.3390/cancers14194705. PMID 36230628
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org